CLINICAL TRIAL: NCT04273646
Title: Clinical Study of Human Umbilical Cord Mesenchymal Stem Cells in the Treatment of Severe COVID-19
Brief Title: Study of Human Umbilical Cord Mesenchymal Stem Cells in the Treatment of Severe COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Wuhan Hamilton Bio-technology Co., Ltd, China. (Unknown)
Responsible Party: Principal Investigator, Yang Jin, Principle Investigator, Clinical Professor of Department of Respiratory and Critical Care Medicine,, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202001
Record Dates: First submitted 2020-02-14; First posted 2020-02-18 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: 2019 Novel Coronavirus Pneumonia; COVID-19
Keywords: 2019 Novel Coronavirus Pneumonia; Safety; Efficiency; Cell Therapy; UC-MSCs
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UC-MSCs Treatment Group (Experimental): Conventional treatment plus UC-MSCs:
  Participants will receive conventional treatment plus 4 times of UC-MSCs(0.5*10E6 UC-MSCs/kg body weight intravenously at Day 1，Day 3，Day 5，Day7).
  Interventions: Biological: UC-MSCs
- Conventional Control Group (Placebo Comparator): Conventional treatment plus Placebo:
  Without UC-MSCs Therapy but conventional treatment should be received. Participants will receive conventional treatment plus 4 times of Placebo intravenously at Day 1，Day 3，Day 5，Day7).
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: UC-MSCs — 4 times of UC-MSCs(0.5*10E6 UC-MSCs/kg body weight intravenously at Day 1, Day 3, Day 5, Day 7).
  Arms: UC-MSCs Treatment Group
Drug: Placebo — 4 times of cell-free stem cell suspension (saline containing 1% human albumin) intravenously at Day 1, Day 3, Day 5, Day 7).
  Arms: Conventional Control Group

SUMMARY:
The novel coronavirus pneumonia is a kind of new emerging respiratory infectious disease, characterized by fever, dry cough, and chest tightness, and caused by the infection of the 2019 novel coronavirus (2019-nCoV). In severe cases, there will be rapid respiratory system failure. The novel coronavirus pneumonia is extremely contagious and the disease progresses rapidly. It has become a urgent and serious public health event that threatens human life and health globally. Among them, severe pneumonia caused by novel coronavirus is characterized by extensive acute inflammation of the lungs and the patient is critically ill. At present, there is no effective treatment in clinical practice.Most of them should receive supportive care to help relieve symptoms. For severe cases, treatment should include care to support vital organ functions. This clinical trial is to inspect the safety and efficiency of Human Umbilical Cord Mesenchymal Stem Cells (UC-MSCs) therapy for severe pneumonia patients infected with 2019-nCoV.

DETAILED DESCRIPTION:
Since December 2019, Wuhan has successively found multiple cases of patients with pneumonia infected by a novel coronavirus. With the spread of the epidemic, other cases in China and abroad have also found such cases. As of 24:00 on February 1, 2020, a total of 14,380 confirmed cases were reported in China, of which there were 2110 severe cases and 304 death cases. At present, there is no effective treatment for pneumonia in the clinic against new coronavirus infection, especially severe and critical cases. Therefore, it is of great significance to explore more active and effective therapeutic approach to severe pneumonia patients infected with 2019-nCoV.

Human and animal studies have shown that after infection with coronavirus, the rapid replication of the virus in the body and the subsequent inflammatory response cause damage to alveolar epithelial cells and capillary endothelial cells, causing diffuse interstitial and alveolar edema, and pulmonary function. Impaired, leading to acute hypoxic respiratory insufficiency. The National Health and Medical Commission recently released the "New Coronavirus Infected Pneumonia Diagnosis and Treatment Plan (Trial Version 5)", which pointed out that the new type of coronavirus severe pneumonia usually has difficulty breathing after one week, and the severe cases quickly progress to acute respiratory distress syndrome, Septic shock and metabolic acidosis that is difficult to correct. It can be seen that the key to the treatment of new coronavirus severe pneumonia is to inhibit the super-inflammatory immune response caused by the virus, thereby reducing the damage of alveolar epithelial cells and capillary endothelial cells, and then repairing the structure and function of lung tissue.

Mesenchymal stem cells (MSCs) are one of the most studied and important adult stem cells. A large amount of evidence shows that MSCs can migrate to and return to damaged tissues, exert strong anti-inflammatory and immune regulatory functions, promote the regeneration and repair of damaged tissues, resist apoptosis and inhibit tissue fibrosis, and reduce tissue damage. Many studies have shown that the anti-inflammatory effects of MSCs can significantly reduce virus-induced lung injury and mortality in mice. Studies have shown that MSCs can significantly reduce acute lung injury in mice caused by H9N2 and H5N1 viruses by reducing the levels of proinflammatory cytokines and chemokines and reducing the recruitment of inflammatory cells into the lungs. Compared with MSCs from other sources, human umbilical cord-derived MSCs (umbilical cord MSCs, UC-MSCs) have been widely used because of their convenient collection, no ethical controversy, low immunogenicity, fast self-renewal and strong proliferation ability Research on the treatment of various diseases. Early research in this laboratory used UC-MSCs to intervene in endotoxin (LPS) -induced acute lung injury in mice, and confirmed that UC-MSCs can significantly reduce inflammatory cell infiltration in lung tissue, reduce inflammation in lung tissue, and significantly improve lung The structure and function of tissues protect mouse lung tissue from endotoxin-induced damage.

The purpose of this study is to investigate efficiency and safety of UC-MSCs in treating severe pneumonia patients infected with 2019-nCoV. This trial will recruit 48 patients. 24 patients received i.v. transfusion one round (4 times) of 5.0*10E6 cells/kg of UC-MSCs as the treated group, all of them received the conventional treatment. In addition, the equal 24 patients received conventional treatment were used as control group. The respiratory function, pulmonary inflammation, clinical symptoms, pulmonary imaging, side effects, 28-days mortality, immunological characteristics (immune cells, inflammatory factors, etc.) will be evaluated during the 90 days to 96 weeks follow up.

ELIGIBILITY:
Inclusion Criteria:

1. CT image is characteristic of viral pneumonia;
2. 2019-ncov infection (positive nucleic acid test) is confirmed by pathogenic test;
3. In compliance with the 2019-nCoV infection severe pneumonia diagnosis standard (according to the novel coronavirus infection pneumonia diagnosis and treatment program (Trial Implementation Version 5) issued by the National Health and Medical Commission, and WHO 2019 new coronavirus guidelines standards). It is severe if it meets any of the following: (A) Increased breathing rate (≥30 beats / min), difficulty breathing, cyanosis of the lips; (B) When inhaling, means oxygen saturation ≤93%; (C) Partial pressure of arterial oxygen (PaO2) / Fraction of inspired oxygen (FiO2) ≤300 mmHg (1mmHg = 0.133kPa);
4. 18 years old ≤ age ≤ 65 years old, regardless of gender;
5. The patient or legal donor agrees to participate in the study and signs the informed consent.

Exclusion Criteria:

1. Patients with severe allergies or allergies to stem cell preparations and their components;
2. Patients with serious basic diseases that affect survival, including: blood diseases, cachexia, active bleeding, severe malnutrition, etc .;
3. Patients with pulmonary obstructive pneumonia, severe pulmonary interstitial fibrosis, alveolar proteinosis, allergic alveolitis, and other known viral pneumonia or bacterial pneumonia;
4. Continuous use of immunosuppressive agents or organ transplants in the past 6 months;
5. In vitro life support (ECMO, ECCO2R, RRT);
6. Expected deaths within 48 hours, uncontrolled infections;
7. Patients with malignant blood-borne diseases such as HIV or syphilis;
8. Patient with pregnancy, are planning to become pregnant or breastfeeding;
9. Patients with poor compliance and unable to complete the full study;
10. The investigator determines that there may be increased risk of the subject or other conditions that interfere with the clinical trial and the judgment of the results (such as excessive stress, sensitivity or cognitive impairment, etc.);
11. There are other situations that the researchers think are not suitable to participate in this clinical study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-04-20 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2022-02-15 (Estimated)

PRIMARY OUTCOMES:
Pneumonia severity index | From Baseline (0W) to 12 week after treatment
  Evaluation of Pneumonia Improvement
Oxygenation index (PaO2/FiO2) | From Baseline (0W) to 12 week after treatment
  Evaluation of Pneumonia Improvement

SECONDARY OUTCOMES:
Side effects in the UC-MSCs treatment group | From Baseline (0W) to 96 week after treatment
  Incidence of acute and chronic treatment-related adverse events in patients with novel coronavirus severe pneumonia receiving UC-MSCs infusion as assessed.
28-days survival | Day 28
  Marker for efficacy of treatment
Sequential organ failure assessment | Day 28
  Markers of organ function（Score each criterion on a scale of 0 to 4, and the higher the score, the worse the prognosis.）
C-reactive protein | From Baseline (0W) to 12 week after treatment
  Markers of Infection
Procalcitonin | From Baseline (0W) to 12 week after treatment
  Markers of Infection
Lymphocyte count | From Baseline (0W) to 12 week after treatment
  Marker of Immunological function
CD3+, CD4+ and CD8+ T celll count | From Baseline (0W) to 12 week after treatment
  Marker of Immunological function
CD4+/CD8+ratio | From Baseline (0W) to 12 week after treatment
  Marker of Immunological function

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No